**Study Title:** Improving Influenza Vaccination Delivery Across a Health System by the Electronic

Health Records Patient Portal RCT 6

Initial IRB Approval: 12/20/2017

**RCT 6 IRB Approval:** 08/11/2023

Clinical Trials Registration: NCT06062264

# **Brief Summary:**

This trial is taking place in Los Angeles, CA at 21 clinics within the UCLA Health System.

The study design is a 3 arm randomized trial. Patients will be randomized into 1) receiving portal based reminder messages with a video from their PCP encouraging them to receive the influenza vaccine, 2) portal-based reminder messages with an infographic with the image of their PCP encouraging them to receive the influenza vaccine, or 3) the control group. Patients randomized to the intervention arms will receive reminders if they are due for influenza vaccine.

Despite the Advisory Committee on Immunization Practices (ACIP) recommendation in 2010 that all people above 6 months of age should receive an annual flu vaccine, vaccination rates remain low: at 6m-4.9 yrs. (70%), 5-17.9 yrs. (56%), 18-64.9 yrs. (38%), and >65 yrs. (63%). The investigators will assess the effectiveness of MyChart R/R video messages and infographic messages as compared to the standard of care control (Health system messages).

## **Methods and Procedures**

This randomized controlled trial will assess the effectiveness of reminders messages sent to portal users, encouraging influenza vaccination, on increasing influenza vaccination rates within a health system. Patients will be randomized into three groups: 1) one-third of patients will receive reminder messages with a video from their PCP encouraging them to receive the influenza vaccine, 2) one-third will receive reminders with an infographic with information about the influenza vaccine with an image of their PCP, and 3) one-third will receive standard health system messages (standard of care).

Portal-based video messages: Clinicians have been shown to be trusted by their patients, so by sending patients videos that have been recorded by their own primary care physician, we are testing the concept of 'trusted messengers' to improve influenza vaccine uptake.

Portal-based infographic messages: This study arm is also testing the concept of 'trusted messenger' since all infographic messages will also have an image of patients' own primary care physician at the top.

Interventions that apply Behavioral Economics principles in vaccine promotion messaging can increase vaccine receipt. In the physician videos and infographics we will also include language utilizing the concepts endorsing social norms, social good, positive framing, urgency, and planning.

For the primary analysis, the primary outcome will be the patient's end of flu season vaccination status. Intervention effects will be assessed using mixed effects log-binomial models.

The portal-based reminder messages will be sent in October of 2023. Repeat messages will also be sent in late October, and late November to patients who do not receive their influenza vaccines.

**Eligibility**: Our EHR will identify subjects who are eligible for either 1 or 2 influenza vaccinations based on ACIP algorithms (2 are recommended for children <9 years who have not had prior vaccination).

## Inclusion criteria

Inclusion criteria will involve-- all patients over 6 months of age who have made at least 1 visit to the practice within the prior 3 years and who have signed up for MyUCLAhealth (UCLA's portal) and have used the portal at least once within 12 months. Currently this includes 145,684 patients.

- a. Active patient: We selected >1 visit in 3y based on our prior studies and the literature to focus the intervention on active patients; practices do not have a good mechanism to inactivate patients.
- b. Focusing on Portal Users: We can only send portal R/R messages to patients who have signed up for the portal. Since some patients sign up for the portal but never use it we will restrict our inclusion criteria to patients who used the portal within 12m (53% of UCLA patients). This standard has been applied before. We will assess intervention effects for the included population, and also for the entire practice, since the impact of the intervention reflects the extent of portal penetration.

### **Exclusion criteria**

Patients will be excluded if they are not a patient at one of the 49 primary care practices within UCLA's Health System, and/or if they do not meet the above specified requirements for being an active patient or portal user.

## **Main Outcomes and Measures**

Primary Measure: Receipt of >1 influenza vaccine as documented in the EHR which is supplemented electronically by the health system with influenza vaccination data from external sources (e.g., pharmacies).

| Participant Group/Arm | Intervention/Treatment |
|---|---|
| Active Comparator: Portal-Based PCP Video Reminder Message Participants in their arm will receive up to 3 portal-based messages with a video recorded message from their own primary care physician encouraging them to receive the influenza vaccine. | Video recorded by physician encouraging patients to receive influenza vaccine. Sent via the patient portal. |
| Active Comparator: Portal-Based PCP Infographic Reminder Message Participants in their arm will receive up to 3 portal-based messages with an infographic message with an image of their own primary care | Behavioral: Portal-based Infographic Message Infographic with information about the influenza vaccine and an image of the physician. Sent via the patient portal. |

| physician encouraging them to receive the influenza vaccine. |
|---|
| No Intervention: Standard Health<br>System Portal Messages<br>Participants in this arm will only<br>receive standard-of-care health<br>system portal messages, and will not<br>receive study-based messages. |